CLINICAL TRIAL: NCT05286983
Title: Multidimensional Assessment of Infant, Parent and Staff Outcomes During a Family Centered Care Enhancement Project in a Tertiary Neonatal Intensive Care
Brief Title: Multidimensional Assessment of Infant, Parent and Staff Outcomes During a Family Centered Care Enhancement Project
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: University of Ulm (Other)
Responsible Party: Principal Investigator, Dr. Rahel Schuler, Consultant Neonatology, University of Giessen
Other Study IDs: 153/20
Record Dates: First submitted 2022-02-23; First posted 2022-03-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Family Centered Care
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (11):
- K0 - baseline cohort: 45 preterm infants and their parents (average number of patient admissions per 6 months during the last 5 years)
- K1 - 1st intervention cohort: All preterm infants and their parents enrolled during the first 6 months period after completion of the baseline cohort and who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K2 - 2nd intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K3 - 3rd intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K4 - 4th intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K5 - 5th intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K6 - 6th intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K7 - 7th intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K8 - 8th intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K9 - 9th intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)
- K10 - 10th intervention cohort: All preterm infants and their parents enrolled during the 6 months period after the previous 6 months period who are treated according to prespecified Family Centred Care interventions implemented as Potentially Better Practices.
  Interventions: Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs)

INTERVENTIONS:
Behavioral: Family Centred Care (FCC) interventions as potentially better practices (PBPs) — After the previous period, additional Family Centred Care (FCC) elements will be introduced gradually every 6 months, covering staff training, parent education, psychosocial support for families, and last but not least, the neonatal intensive care unit environment.
  The focus group consisting of nurses and healthcare professionals will meet regularly and will decide on new FCC interventions as potentially better practices (PBPs). New additional PBPs will be disseminated into the greater team through workshops, hands-on teaching, displays, etc. Potential PBPs for our department enclose:
  Parent participation on rounds Parent skill self-assessment Parent-to-parent support Regular staff education Improvement of psychosocial support Improvement of neonatal unit surroundings to promote parent-infant-closeness
  Groups: K1 - 1st intervention cohort; K10 - 10th intervention cohort; K2 - 2nd intervention cohort; K3 - 3rd intervention cohort; K4 - 4th intervention cohort; K5 - 5th intervention cohort; K6 - 6th intervention cohort; K7 - 7th intervention cohort; K8 - 8th intervention cohort; K9 - 9th intervention cohort

SUMMARY:
This prospective single centre longitudinal cohort study enrols preterm infants ≤32+0 weeks of gestation and/or birthweight ≤1500g and their parents. Following a baseline period additional Family Centred Care elements are introduced as potentially better practices, these elements focus on four areas: the NICU (Neonatal Intensive Care Unit) environment, staff training, parental education and psychosocial support to the families. The effect of the implementation of additional Family Centred Care elements on infant, parent and staff outcomes are assessed. The parallel data collection enables to study the interrelation between these three important areas of research.

DETAILED DESCRIPTION:
Background: The therapeutic advances and progress in the care for preterm infants have enabled the regular survival of more and more immature infants. However, the high burden of lifelong sequelae following premature delivery constitutes an ongoing challenge and psychomotor disorders and neurobehavioral difficulties persist into adulthood. Regardless of premature delivery, parental mental health and a healthy parent-child relationship were identified as essential prerogatives for normal infant development. Family centered care (FCC) supports preterm infants and their families by respecting the particular developmental, social and emotional needs in the NICU. Due to the large variations in concepts and goals of different FCC initiatives, scientific data on the benefits of FCC for the infant and family outcome are sparse and its effects on the clinical team need to be elaborated.

Methods: This prospective longitudinal single-center cohort study will enroll preterm infants with a gestational length of ≤32+0 weeks and/or a birth weight of ≤1500 g and their parents. After a baseline period, additional FCC elements will be introduced gradually every 6 months, covering staff training, parent education, psychosocial support for families, and last but not least, the neonatal intensive care unit environment. Recruitment will occur over a 5.5-year period, and outcomes will be tracked through periodic follow-up until 24 month of corrected age. Sample size calculation is based on corrected gestational age at discharge as the primary outcome. Secondary outcomes in infants include morbidities and treatment aspects of prematurity such as somatic growth, duration of ventilatory support, and psychomotor development. Parental outcomes relate to success of parenting education and skills, parent-family interaction, parental satisfaction, and mental health with particular emphasis on anxiety, depression, and stress. Staffing issues are addressed with special attention to the job satisfaction item. Quality improvement steps are monitored using the Plan-Do-Study-Act (PDSA) cycle method, and outcome measures address the child, parent, and medical team as they are inextricably linked. Parallel data collection allows for the interrelationship between these three important research areas to be examined.

Discussion: It is scientifically impossible to allocate improvements in outcome measures to individual enhancement steps of FCC that constitutes a continuous change in NICU culture and attitudes covering diverse areas of change. Therefore, our trial is designed to allocate childhood, parental and staff outcome measures during the stepwise changes introduced by a FCC intervention program. But even if no positive outcome measures can be confirmed, the successful execution of our standardized statistical process control method approach is suited to guide quality improvement in future studies in neonatology and beyond.

ELIGIBILITY:
Inclusion Criteria:

* ≤32+0 weeks of gestational age (GA) and/or birthweight ≤1500g
* biparental (or guardian) written informed consent

Exclusion Criteria:

* severe congenital anomalies (e.g. cyanotic heart disease, severe lung hypoplasia, congenital diaphragmatic hernia)
* decision not to provide full life support
* decision for palliative care before study entry
* parents with severe psychiatric disease

Ages: 1 Minute to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of inborn and outborn preterm infants of ≤32+0 weeks of gestational age (GA) and/or birthweight ≤1500g who are admitted to the Level 3 NICU and their parents
Sampling Method: Probability Sample
Enrollment: 495 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 5.5years
  Length of hospital stay measured by corrected gestational age at discharge

SECONDARY OUTCOMES:
Key neonatal morbidities | 5.5years
  Number of Participants with Bronchopulmonary Dysplasia (BPD), Number of Participants with Intraventricular Hemorrhage (IVH) Grade III-IV, Number of Participants with Periventricular Leucomalacia (PVL), Number of Participants with Necrotizing Enterocolitis (NEC) stage 2 or stage 3, Number of Participants with Retinopathia of Prematurity (ROP) stage 3 or greater or treatment
Weight gain | 5.5years
  weight gain (g/kg/d) from admission to 36+0/40+0 weeks (corrected age)
Weight Z-Score | 5.5years
  Z- Scores for weight at 36+0, 40+0, 3, 12 and 24 months (corrected age)
Weight | 5.5years
  Weight in Gram at 36+0, 40+0, 3, 12 and 24 months (corrected age)
Length Z-Score | 5.5years
  Z- Scores for length at 36+0, 40+0, 3, 12 and 24 months (corrected age)
Length | 5.5years
  Length in cm at 36+0, 40+0, 3, 12 and 24 months (corrected age)
Head Circumference Z-Score | 5.5years
  Z- Scores for head circumference at 36+0, 40+0, 3, 12 and 24 months (corrected age)
Head Circumference | 5.5years
  Head circumference in cm at 36+0, 40+0, 3, 12 and 24 months (corrected age)
Full enteral feeds | 5.5 years
  Day of Life (DOL) of achievement of full enteral feeds defined as 150ml/kg/d for 3 consecutive days
Length of tube feeding | 5.5 years
  corrected gestational age at removal of nasogastric tube
First Breastmilk Feed | 5.5years
  DOL (Day of Life) with first breast milk feed
Breastmilk Nutrition | 5.5years
  Breastmilk proportion within Day of Life (DOL) 1-14
Fully Breastfed | 5.5years
  DOL when infant is fed only with breast milk
Breastfeeding at Discharge | 5.5years
  Breast milk proportion at discharge
Mechanical ventilation | 5.5years
  Gestational age (GA) at end of respiratory support: Continuous Positive Airway Pressure (CPAP)/ Highflow Nasal Cannula (HFNC)/ oxygen supplementation
End of parenteral nutrition (PN) | 5.5years
  DOL of end of PN
Family room | 5.5years
  cGA at move-in with mother or father into a family room
Neurodevelopment at 12 months corrected age | 7.5years
  Neurodevelopment measured with Neuropsychological Developmental Screening, Score 0-15, higher scores indicating better neurodevelopment
Neurodevelopmental outcome at 24 months corrected age | 7.5years
  Neurodevelopmental outcome measured with Bayley Scales of Infant Development, German Version, 3rd Edition (mean 100; Standard Deviation 15, higher Scores indicating better neurodevelopment)
Motor Developmental outcome at 24 months corrected age | 7.5years
  Gross Motor Function Classification System (GMFCS), Grade I-V, higher Grade indicating worse motor outcome
Parental Anxiety | 5.5years
  Parental Anxiety, measured with the German version of the Hospital and Anxiety and Depression Scale (HADS-D) within the first 10 days after birth, after 4 weeks, at discharge, at 3, 12 and 24 months (corrected age of the preterm infant), Score 0-21; higher scores indicating more anxiety
Parental Depression | 5.5years
  Parental Depression measured with the German version of the Hospital and Anxiety and Depression Scale (HADS-D) within the first 10 days after birth, after 4 weeks, at discharge, at 3, 12 and 24 months (corrected age of the preterm infant), Score 0-21, higher scores indicating more depression
Parental Stress | 5.5years
  Parental Stress measured with the Parenting Stress Index (PSI), German Version (Eltern-Belastungs-Inventar, EBI) within the first 10 days after birth, after 4 weeks, at discharge, at 3, 12 and 24 months (corrected age of the preterm infant); Score 0-100, higher score indicating more stress
Parental Satisfaction | 5.5years
  Measured with a newly designed Questionnaire focussing on Neonatal Intensive Care Surroundings, Visiting Hours, Medical Care and communication
Parental Skills | 5.5years
  Self assessed with a Questionnaire
Parental Visiting Hours | 5.5years
  Time spent with the infant. Measured seperately for mothers and fathers throughout hospital stay
Degree of Family Centred Care | 5.5years
  Self Assessment Questionnaire (Institute for Family Centred Care) by staff members
Staff satisfaction | 5.5years
  Self assessment (Copenhagen Psychosocial Questionnaire, COPSQ) by staff members
Kangarooing time | 5.5yrs
  Time spent kangarooing with the infant. Measured separately for mothers and fathers throughout the NICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Rahel Schuler, Principal Investigator — Department of General Pediatrics and Neonatology, Justus- Liebig- University, Giessen, Germany
Locations (2):
- Germany (2):
  - Mihatsch Walter, Ulm, Baden-Wurttemberg
  - Department of General Pediatrics and Neonatology, Justus- Liebig- University, Feulgenstrasse 12, D-35392 Giessen, Germany, Giessen, Hesse

REFERENCES:
- [Background] Schuler R, Ehrhardt H, Mihatsch WA. Safety and Parental Satisfaction With Early Discharge of Preterm Infants on Nasogastric Tube Feeding and Outpatient Clinic Follow-Up. Front Pediatr. 2020 Aug 25;8:505. doi: 10.3389/fped.2020.00505. eCollection 2020. PMID 32984217
- [Derived] Schuler R, Woitschitzky L, Eiben C, Beck J, Jagers A, Windhorst A, Kampschulte B, Petzinger J, Waitz M, Kilsdonk MOR, Neubauer BA, Zimmer KP, Ehrhardt H, Brosig B, Mihatsch WA. Multidimensional assessment of infant, parent and staff outcomes during a family centered care enhancement project in a tertiary neonatal intensive care unit: study protocol of a longitudinal cohort study. BMC Pediatr. 2023 Jul 7;23(1):344. doi: 10.1186/s12887-023-04165-0. PMID 37420180